CLINICAL TRIAL: NCT06819852
Title: Skipping the Hospital: Acute Hospital Care at Home for People Living With Dementia
Brief Title: Acute Hospital Care at Home for People Living With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, David Levine, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P000002; R01AG082771-01A1 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Emergency Department Visit; Home Care Services; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data collectors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Acute care at a brick-and-mortar hospital.
  Interventions: Other: Standard medical treatment
- Acute hospital care at home (Experimental): Home visit for a serious illness conversation. Acute illness evaluation on demand. Acute hospital care at home as needed.
  Interventions: Other: Acute hospital care at home

INTERVENTIONS:
Other: Acute hospital care at home — Home visit for a serious illness conversation. Acute illness evaluation on demand. Acute hospital care at home as needed.
  Arms: Acute hospital care at home
Other: Standard medical treatment — Standard acute and emergency care delivered in a brick-and-mortar hospital setting.
  Arms: Usual care

SUMMARY:
The investigators will perform a parallel-group multicenter randomized controlled trial of a 1-year pre-enrolled acute hospital care at home intervention vs usual care for people living with dementia. Patients will be randomized only after eligibility determination and after the family caregiver agrees to enroll; people living with dementia will assent when able. Patients will be allocated in a concealed fashion to the control and intervention groups in randomly selected block sizes of 4 or 6 in 4 strata reflecting their functional status (activities of daily living: 0, 1, 2-3, 4-6). Although family and clinicians cannot be blinded, the investigators will blind the data collectors and assessors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate or severe dementia (as ascertained by the Quick Dementia Rating System; QDRS)
* Resides in a private or assisted living residence with or nearby (<15min travel time) to a family caregiver
* Resides within the Mass General Brigham (MGB) home hospital catchment area
* Has had at least 1 hospitalization in the last 12 months.

Exclusion Criteria:

* No functioning utilities, such as no working heat (October-April), no running water, or no electricity.
* Resides in skilled nursing facility
* Resides in group home
* Domestic violence screen positive
* In police custody
* Family caregiver unable to initiate or maintain communication with care team
* End-stage renal disease on hemodialysis
* On methadone requiring daily pickup of medication
* Active substance use disorder, without functioning treatment plan
* Psychiatric diagnosis that would prohibit successful home hospital care
* Acute delirium without explanation or without the ability to manage at home
* Patients with cancer requiring consistent hospital-based treatments
* Cannot ambulate to bedside commode with assistance present in the home (if different from baseline), unless home-based aides are available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of days at home | Discharge to 30-days post discharge, up to 30 days
  Sum of the number of days spent at home within the 30-days after an acute care episode

SECONDARY OUTCOMES:
30-day unplanned readmission or mortality | Discharge to 30-days post discharge, up to 30 days
  Percentage of unplanned readmissions or mortality
Delirium | Date of admission to date of discharge, estimated 5 days
  Percentage of days experiencing delirium while receiving acute care using the short confusion assessment method.
Health-related quality of life | From enrollment for the period of one year
  Absolute change of health-related quality of life over the year through the dementia quality of life survey (DEMQOL), or for patients unable to complete the survey, its proxy version (DEMQOL-Proxy).
Physical activity | Date of admission to date of discharge, estimated 5 days
  Percent of time sedentary as measured by patch monitoring system.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No